Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

Are you participating in any other research studies? \_\_\_\_\_ Yes \_\_\_\_\_No

#### **PURPOSE OF RESEARCH**

You are invited to participate in a research study of preventing lymphedema with the Lymphatic Microsurgical Preventative Healing Approach (LYMPHA). We hope to learn if there is a role for this low risk procedure in preventing lymphedema in those undergoing surgery for breast cancer. You were selected as a possible participant in this study because you will be undergoing surgery for breast cancer that included axillary lymph node dissection and increases your risk of lymphedema.

If you decide to terminate your participation in this study, you should notify Dr. Dung Nguyen at 650-498-6004. Mailing address: 900 Blake Wilbur Dr f1, Palo Alto, CA 94304

This research study is looking for 80 with breast cancer. Enrollment will occur at Stanford University. Stanford University expects to enroll 80 research study participants.

## **VOLUNTARY PARTICIPATION**

Your participation in this study is entirely voluntary. Your decision not to participate will not have any negative effect on you or your medical care. You can decide to participate now, but withdraw your consent later and stop being in the study without any loss of benefits or medical care to which you are entitled.

#### **DURATION OF STUDY INVOLVEMENT**

This research study is expected to take approximately 2 years with 1 year of follow-up minimum for every patient.

#### **PROCEDURES**

This is a randomized control trial, meaning that half of participants will receive the procedure and the other half of the participants will not. This decision is made at random. If you choose to participate, you will be randomly assigned to


Participant ID:



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

either the group that will receive the LYMPHA procedure, or the group that will not. If you are in the group that will receive the procedure, Dr. Dung Nguyen and her research study staff will perform the LYMPHA procedure at the time of your cancer operation.

The LYMPHA procedure include attaching veins to lymphatics in the axilla where the lymphatics would normally be destroyed and not repaired by the axillary dissection. This is the standard of care for preventing lymphedema. Approximately 45 minutes to 1 hours will be added to the procedure time. There is no additional risk associated with this addition.

All patients (in both groups) will undergo an initial study evaluation to establish the pre-operative baseline and to determine eligibility for randomization. Each of the baseline measures will be repeated at 3-month intervals over the 12 months of enrollment in the study. These include lymphography, limb volume measurements, skin thickness measurements, bioimpedance spectrosocpy, and quality-of-life assessment.

## Women of Childbearing Potential

If you are a woman who is able to become pregnant, it is expected that you will use an effective method of birth control to prevent exposing a fetus to a potentially dangerous agent with unknown risk. If you are pregnant or currently breast feeding, you may not participate in this study. You understand that if you are pregnant, if you become pregnant, or if you are breast-feeding during this study, you or your child may be exposed to an unknown risk.

To confirm to the extent medically possible that you are not pregnant, you agree choose to have a pregnancy test done before beginning this research study or to begin the study after the onset of your next menstrual period. You must agree to avoid sexual intercourse or use a birth control method judged to be effective by the investigator and which will not interfere with the proposed investigation. You must accept the risk that pregnancy could still result despite the responsible use of reliable method of birth control. You agree to notify the investigator as soon as possible of any failure of proper use of your birth control method, or if you become pregnant, either of which may result in your being withdrawn from the study.

## PARTICIPANT RESPONSIBILITIES


Participant ID:



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

As a participant, your responsibilities include:

- Follow the instructions of the Protocol Director and study staff.
- Keep your study appointments. If it is necessary to miss an appointment, please contact the Protocol Director or research study staff to reschedule as soon as you know you will miss the appointment.
- Tell the Protocol Director or research study staff about any side effects, doctor visits, or hospitalizations that you may have.
- Tell the Protocol Director or research staff if you believe you might be pregnant.
- Complete your questionnaires as instructed.
- Ask questions as you think of them.
- Tell the Protocol Director or research staff if you change your mind about staying in the study.

#### WITHDRAWAL FROM STUDY

If you first agree to participate and then you change your mind, you are free to withdraw your consent and discontinue your participation at any time. Your decision will not affect your ability to receive medical care for your disease and you will not lose any benefits to which you would otherwise be entitled.

If you decide to withdraw your consent to participate in this study, you should notify Dr. Dung Nguyen at 650-498-6004.

If you withdraw from the study:

- There are no anticipated consequence from withdrawing from the study
- If you wish to withdrawal from the study, please contact the program director and you will be withdrawn

The Protocol Director may also withdraw you from the study, without your consent for one or more of the following reasons

Failure to follow the instructions of the Protocol Director and study staff.

- The Protocol Director decides that continuing your participation could be harmful to you.
- Pregnancy



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022


NCT: NCT05366699

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

- You need treatment not allowed in the study.
- The study is cancelled.
- Other administrative reasons.
- Unanticipated circumstances.

## POSSIBLE RISKS, DISCOMFORTS, AND INCONVENIENCES

There are risks, discomforts, and inconveniences associated with any research study. These deserve careful thought. You should talk with the Protocol Director if you have any questions.

The LYMPHA procedure is a normal part of the clinical treatment of this condition. Patients in both the treated and untreated groups are subject to the baseline risk of surgical intervention, including but not limited to bleeding, infection, scar, injury to surrounding structures, risks of anesthesia, and need for further surgery.

Addition of the LYMPHA procedure adds time to the overall operation, approximately 45 minutes to 1 hour.

The study also involves frequent follow up and the inconvenience of traveling to these appointments.

The procedures in this study may involve risks to the subject which are currently unforeseeable.

#### **POTENTIAL BENEFITS**

The LYMPHA procedure may be reasonably expected to decrease your risk of developing lymphedema. We cannot and do not guarantee or promise that you will receive any benefits from this study.

#### **ALTERNATIVES**

The alternative is to not participate. If lymphedema develops later on, at that time there are a number of non-surgical options (compression stockings, therapeutic massage) and surgical therapies available. However, these therapies are typically not curative.

## **PARTICIPANT'S RIGHTS**


Participant ID:

NCT: NCT05366699



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

You should not feel obligated to agree to participate. Your questions should be answered clearly and to your satisfaction. If you decide not to participate, tell the Protocol Director.

You will be told of any important new information that is learned during the course of this research study, which might affect your condition or your willingness to continue participation in this study.

## ClinicalTrials.gov

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## **CONFIDENTIALITY**

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed except as authorized by you or as required by law. However, there is always some risk that even de-identified information might be re-identified.

Patient information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction. Identifiers might be removed from identifiable private information and/or identifiable specimens and, after such removal, the information and/or specimens could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you.

CTI ID) (

IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022


Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

# **Authorization To Use Your Health Information For Research Purposes**

Because information about you and your health is personal and private, it generally cannot be used in this research study without your written authorization. If you sign this form, it will provide that authorization. The form is intended to inform you about how your health information will be used or disclosed in the study. Your information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing it.

## What is the purpose of this research study and how will my health information be utilized in the study?

Lymphedema is a progressive and debilitating disease that significantly affects quality of life. Current therapeutic options for lymphedema are less than optimal. The purpose of this study is to further define the role of the LYMPHA procedure in preventing lymphedema. Your health information will de-identified and used to determine the utility of the LYMPHA procedure. If appropriate the de-identified results of our study will be published.

## Do I have to sign this authorization form?

You do not have to sign this authorization form. But if you do not, you will not be able to participate in this research study, including receiving any research-related treatment. Signing the form is not a condition for receiving any medical care outside the study.

## If I sign, can I revoke it or withdraw from the research later?

If you decide to participate, you are free to withdraw your authorization regarding the use and disclosure of your health information (and to discontinue any other participation in the study) at any time. After any revocation, your health information will no longer be used or disclosed in the study, except to the extent that

Participant ID:

NCT: NCT05366699



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

the law allows us to continue using your information (e.g., necessary to maintain integrity of research). If you wish to revoke your authorization for the research use or disclosure of your health information in this study, you must call or write: Dr. Dung Nguyen at 650-498-6004, 900 Blake Wilbur Dr f1, Palo Alto, CA 94304.

## What Personal Information Will Be Obtained, Used or Disclosed?

Your health information related to this study, may be used or disclosed in connection with this research study, including, but not limited to, your demographics, medical history, cancer history, surveys your complete, and data collected on the operating limb (limb volume, skin thickness, lymphography, and edema content).

## Who May Use or Disclose the Information?

The following parties are authorized to use and/or disclose your health information in connection with this research study:

- The Protocol Director Dr. Dung Nguyen
- The Stanford University Administrative Panel on Human Subjects in Medical Research and any other unit of Stanford University as necessary
- Research Staff

## Who May Receive or Use the Information?

The parties listed in the preceding paragraph may disclose your health information to the following persons and organizations for their use in connection with this research study:

 The Office for Human Research Protections in the U.S. Department of Health and Human Services

Your information may be re-disclosed by the recipients described above, if they are not required by law to protect the privacy of the information.

Participant ID:

NCT: NCT05366699



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

STUDY

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

## When will my authorization expire?

Your authorization for the use and/or disclosure of your health information will end in February 28, 2050 or when the research project ends, whichever is earlier.

## Will access to my medical record be limited during the study?

To maintain the integrity of this research study, you may not have access to any health information developed as part of this study until it is completed. At that point, you would have access to such health information if it was used to make a medical or billing decision about you (e.g., if included in your official medical record).

| Signature of Adult Participant | <br>Date |
|---|---|
| Print Name of Adult Participant | |
| Signature of Legally Authorized Representative (LAR) (e.g., parent, guardian or conservator) | Date |
| Print Name of LAR | |
| LAR's Authority to Act for Participant (e.g., parent, quardian or conservator) | |






IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

## **FINANCIAL CONSIDERATIONS**

## Costs

There is no cost to you for participating in this study, other than basic expenses like transportation and the personal time it will take to come to all of the study visits.

**Compensation** 

Participants will not be paid

## **COMPENSATION for Research-Related Injury**

All forms of medical diagnosis and treatment — whether routine or experimental — involve some risk of injury. In spite of all precautions, you might develop medical complications from participating in this study. If such complications arise, the Protocol Director and the research study staff will assist you in obtaining appropriate medical treatment. In the event that you have an injury or illness that is directly caused by your participation in this study, reimbursement for all related costs of care first will be sought from your insurer, managed care plan, or other benefits program. You will be responsible for any associated co-payments or deductibles as required by your insurance.

If costs of care related to such an injury are not covered by your insurer, managed care plan or other benefits program, you may be responsible for these costs. If you are unable to pay for such costs, the Protocol Director will assist you in applying for supplemental benefits and explain how to apply for patient financial assistance from the hospital.

You do not waive any liability rights for personal injury by signing this form.

#### CONTACT INFORMATION

Questions, Concerns, or Complaints: If you have any questions, concerns or complaints about this research study, its procedures, risks and benefits, or alternative courses of treatment, you should ask the Protocol Director, Dr. Dung Nguyen You may contact her now or later at 650-498-6004.

Injury Notification: If you feel you have been hurt by being a part of this study, please contact the Protocol Director, Dr. Dung Nguyen at 650-498-6004.


Participant ID:

NCT: NCT05366699



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at (650)-723-5244 or toll free at 1-866-680-2906. You can also write to the Stanford IRB, Stanford University, 1705 El Camino Real, Palo Alto, CA 94306.

Appointment Contact: If you need to change your appointment, please contact the Stanford Women's Cancer Center at 650-498-6004.

## **EXPERIMENTAL SUBJECT'S BILL OF RIGHTS**

As a research participant you have the following rights. These rights include but are not limited to the participant's right to:

- be informed of the nature and purpose of the experiment;
- be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized;
- be given a description of any attendant discomforts and risks reasonably to be expected;
- be given an explanation of any benefits to the subject reasonably to be expected, if applicable;
- be given a disclosure of any appropriate alternatives, drugs or devices that might be advantageous to the subject, their relative risks and benefits;
- be informed of the avenues of medical treatment, if any available to the subject after the experiment if complications should arise;
- be given an opportunity to ask questions concerning the experiment or the procedures involved;
- be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation without prejudice;
- be given a copy of the signed and dated consent form; and
- be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion or undue influence on the subject's decision.

IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022


Protocol Director: Dung Nguyen MD

Approval Date: June 15, 2021 Expiration Date: June 15, 2022

IRB Use Only

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after Axillary Lymphadenectomy

| Signing your name means you agree to be in taging a copy of this signed and dated consent form. | this study a | and that you will receive |
|---|---|---|
| Signature of Adult Participant | | Date |
| Print Name of Adult Participant | | |
| Signature of Legally Authorized Representative (e.g., parent, guardian or conservator) | e (LAR) | <br>Date |
| Print Name of LAR | | |
| LAR's Authority to Act for Participant (e.g., parent, guardian or conservator) | | |
| Signature of Person Obtaining Consent | | <br>Date |
| Print Name of Person Obtaining Consent | | |
| The following witness line is to be signed only if th form and accompanied by a short form foreign lan | | |
| Signature of Witness | _ | <br>Date |
| Print Name of Witness | ) | |



rage 11 of 12

Protocol Director: Dung Nguyen MD

Protocol Title: A Randomized Clinical Trial of the LYMPHA procedure for the Prevention of Lymphedema after

Axillary Lymphadenectomy

(e.g., staff, translator/interpreter, family member)

- Translated short form must be signed and dated by both the participant (or their LAR) AND the witness.
- The English consent form (referred to as the "Summary Form" in the regulations):
  - Must be signed by the witness AND the Person Obtaining Consent (POC).
  - The non-English speaking participant/LAR does not sign the English consent.
  - The non-English speaking participant/LAR should not sign the HIPAA participant line
  - If the participant or the LAR is non-English speaking, the Person Obtaining Consent (POC) must ensure that 1) the LAR's Description of Authority is completed and 2) that any questions or options presented by the consent form are documented and initialed by the POC on the Summary Form, per the participant's wishes, as they are understood during the consent process.

Participant ID:

NCT: NCT05366699



IRB Use Only

Approval Date: June 15, 2021 Expiration Date: June 15, 2022